CLINICAL TRIAL: NCT03450447
Title: Outcomes of a Novel Treatment Decision of Patients With Superficial Esophageal Carcinoma Synchronously Associated With Head and Neck Cancer
Brief Title: Outcomes of A Novel Treatment Decision of Patients With Esophageal and Head and Neck Carcinoma Synchronously
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yanqing Li (Other)
Responsible Party: Sponsor-Investigator, Yanqing Li, professor, chief of gastrointestinal department of Qilu hospital of Shandong University, Shandong University
Organization: Shandong University (Other)
Other Study IDs: 2018SDU-QILU-G02
Record Dates: First submitted 2018-02-10; First posted 2018-03-01 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Head and Neck Cancer; Esophageal Cancer Stage
Keywords: Head and Neck Cancer; Esophageal Cancer; endoscopic submucosal dissection; quality of life; median survival time
MeSH Terms: conditions — Head and Neck Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — histopathology of esophageal endoscopic submucosal dissection specimen histopathology of surgical specimen of head and neck
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To summarise the outcomes of a treatment decision of patients with superficial esophageal carcinoma synchronously associated with head and neck cancer, that is endoscopic treatment for the superficial esophageal carcinoma plus surgery of the head and neck carcinoma.

DETAILED DESCRIPTION:
As a same risk factor, such as heavy drinking and smoking, patients with head and ncek carcinoma are always suffering from synchronous esophageal squamous cell carcinoma. Previous studies illustrated that many patients with multiple esophageal lesions of early stage. In clinical practice, those patients are treated by extensive surgical resection of total pharyngo-laryngo-esophagectomy plus free jejunum interposition or gastric tube, then followed by chemoradiotherapy as standard treatment, resulting in a low quality of life for the patients, and due to the above mentioned disadvantages, many patients with synchronous superficial esophageal squamous cell carcinoma and head and neck carcinoma refused the surgery treatment. Our aims is to summarize the the outcomes of endoscopic treatment for the superficial esophageal carcinoma plus surgery of head and neck carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with head and ncek carcinoma associated with synchronous superficial esophageal squamous cell carcinoma.
2. Patients agree to be treated with esophageal endoscopic submucosal dissection firstly, then accept surgery of head and neck carcinoma.

Exclusion Criteria:

1. Patients refuse a endoscopic submucosal dissection or surgery.
2. Patients with sever systemic disease, such as sever cardiopulmonary disease, renal failure and impaired blood coagulation.
3. Obstruction of the pharynx leading to a failure of insertion of endoscopy.
4. Patients with an advanced esophageal carcinoma evaluated by endoscopy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with head and ncek carcinoma and synchronous superficial esophageal squamous cell carcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-03-10 (Estimated); Primary Completion 2020-02-07 (Estimated); Study Completion 2020-05-07 (Estimated)

PRIMARY OUTCOMES:
The first day of food intake of enrolled patients | An average of 1week
  The first day of food intake after surgery of the head and neck carcinoma

SECONDARY OUTCOMES:
The relapse rate of the enrolled patients | an average of 2 years
  the relapse rate of esophageal cancer or head and neck carcinoma respectively of the enrolled patients.
The hospital stay of enrolled patients | An average of 1 month.
  The total hospital stay during the first hospitalization of the enrolled patients
The incidence of stenosis | an average of 2 years
  The average interval of the stenosis
The severity of stenosis | an average of 2 years
  The average diameter of the stenosis

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, Study Director — Department of Gastroenterology, Qilu Hospital, Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
all the clinical features of the patient are available to all the researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: before the start of the study